CLINICAL TRIAL: NCT03854097
Title: Mechanistic Insights Into Changes in Blood Flow Following Application of Intermittent Negative Pressure
Brief Title: Effect of Intermittent Pressure in Patients With PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-014-18
Record Dates: First submitted 2019-02-19; First posted 2019-02-26 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active PAD group (Experimental): -40mmHg of Intermittent Negative Pressure (INP) for 4-8 weeks.
  Interventions: Device: Active Intermittent Negative Pressure (INP)
- Placebo PAD group (Experimental): -10mmHg of Intermittent Negative Pressure (INP) for 4-8 weeks.
  Interventions: Device: Placebo Intermittent Negative Pressure (INP)
- Healthy Volunteers (Experimental): -40 mmHg of Intermittent Negative Pressure (INP) for 5 days
  Interventions: Device: Active Intermittent Negative Pressure (INP)

INTERVENTIONS:
Device: Active Intermittent Negative Pressure (INP) — Application of -40mmHg negative pressure on the lower limb
  Arms: Active PAD group; Healthy Volunteers
Device: Placebo Intermittent Negative Pressure (INP) — Application of -10mmHg negative pressure on the lower limb
  Arms: Placebo PAD group

SUMMARY:
The study will evaluate the effect of intermittent negative pressure (INP) on peripheral arterial disease (PAD) patient vascular function and blood flow. Patients will be given either -40mmHg INP or -10mmHg INP which will act as a placebo. Healthy volunteers will be given -40mmHg INP to evaluate changes in vascular function and blood flow with INP in healthy physiology.

DETAILED DESCRIPTION:
Atherosclerosis occurs when blood supply to the lower limbs is restricted upon accumulation of fat in the arteries. Atheroslerosis in the lower limbs is termed peripheral arterial disease (PAD). The initial symptom is pain in the lower limbs followed by ulceration and gangrene. The literature has indicated that intermittent negative pressure (INP) can be used to reduce pain and facilitate wound healing. INP is a non-invasive technique that aims to increase arterial and skin blood flow in lower limbs and foot. This study aims to investigate the underlying mechanisms that are involved in changes in blood flow following application of INP. The Flow-Ox 'boot' will be used to apply INP for periods ranging from 4-8 weeks, for an hour twice per day, to the lower limb to determine the effects of INP on vascular function and blood flow. Specifically, vascular tests such as assessments of endothelial function, arterial stiffness, ankle-brachial pressure index (ABPI) and blood borne metabolic and inflammatory markers will be performed before and after INP application. A pain chart will be employed before and after INP application to determine whether there is any change in perception of pain felt by individuals who suffer from pain associated with lower limb arterial disease.

ELIGIBILITY:
Inclusion Criteria

PAD Patients:

* Age ≥ 18 years
* Attending vascular outpatient clinics or admitted in ward with PAD.
* ABPI <0.9

Healthy Volunteers:

* Age ≥ 18 years
* No current or previous significant cardiovascular illness
* Able to give written informed consent

Exclusion criteria

PAD Patients:

* Unable to give written informed consent
* Patients with deep venous thrombosis
* Pregnant women

Healthy Volunteers:

* Positive medical history of: Vascular diseases such as PAD, stroke, IHD, hypertension... etc.
* Haematological conditions such as hypercoagulability, deep venous thrombosis... etc.,
* Alcohol excess
* Unable to give written informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Change in microvascular blood flow | Baseline, 1 day and 4-8 weeks
  Microvascular blood flow measurement in foot using laser Dopper imaging.
Change in microvascular endothelial function | Baseline, 1 day and 4-8 weeks
  Peak blood perfusion response to acetylcholine (ACh) delivered by iontophoresis will be measured using a laser Doppler imager.
Change in arterial stiffness | Baseline, 1 day and 4-8 weeks
  Brachial pulse wave analysis (PWA) augmentation index (Ax) and carotid-femoral pulse wave velocity (m/s) (PWV) as an indication of arterial stiffness.
Change in macrovascular endothelial function | Baseline, 1 day and 4-8 weeks
  Brachial endothelial function measured as change in brachial blood vessel diameter (%) upon shear stress.

SECONDARY OUTCOMES:
Change in pain score | Baseline, 1 day and 4-8 weeks
  Self-scoring of pain felt by patient on a visual analogue scale with 0 being no pain at all to 10 being the worst pain ever felt.
Change in concentration of blood borne inflammatory and oxidative stress biomarkers | Baseline, 1 day and 4-8 weeks
  Concentration of inflammatory and oxidative stress markers of endothelial activation/damage (including IL-1a, IL-6, IL-10, TNF-a, CRP, E-selectin and sICAM-1) measured in serum and plasma collected from patient blood samples.
Change in Ankle-Brachial Pressure Index (ABPI) | Baseline, 1 day and 4-8 weeks
  Brachial systolic pressure and ankle (dorsalis pedis) systolic pressure (mmHg) measured using Doppler probe. ABPI calculated as ankle systolic pressure divided by brachial systolic pressure.
  ABPI <0.9 = PAD, ABPI =>1.0 Normal.

CONTACTS AND LOCATIONS:
Overall Officials: Jody McIntosh, Principal Investigator — PhD student
Locations (1):
- School of Medicine, University of Dundee, Ninewells Hospital & Medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03854097/Prot_SAP_001.pdf